CLINICAL TRIAL: NCT02720900
Title: Effect of a Prebiotic (B-GOS) Supplementation on Microbiota and Gastrointestinal (GI) Symptoms in Children With Autism Spectrum Disorders (ASD)
Brief Title: Prebiotic Intervention for Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clasado Limited (Industry)
Collaborators: University of Reading (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASD2015
Record Dates: First submitted 2015-11-10; First posted 2016-03-28 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — maltodextrin; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maltodextrin (Placebo Comparator): powder, 1.8g/day
  Interventions: Dietary Supplement: Maltodextrin
- B-GOS (Active Comparator): powder, 1.8g/day
  Interventions: Dietary Supplement: B-GOS

INTERVENTIONS:
Dietary Supplement: B-GOS — 1.8 g/day for 6 weeks
  Other Names: Bimuno
  Arms: B-GOS
Dietary Supplement: Maltodextrin — 1.8 g/day for 6 weeks
  Other Names: Corn Starch
  Arms: Maltodextrin

SUMMARY:
The purpose of this study is to determine the effect of a prebiotic (BGOS) on gut microbiota and metabolites in children with autism spectrum disorders.

DETAILED DESCRIPTION:
Children with ASD have a higher incidence of dietary and/or bowel problems than typically developing children. it has been postulated that imbalances in the gut bacteria and/or metabolites present in the gut may be a contributing factor to these symptoms, with potentially bad (toxin-producing) bacteria colonising the gut. Certain carbohydrates (so-called 'prebiotics') are not digested by the human gut and they provide food for beneficial bacteria and thus they improve the composition by preventing the growth of bad bacteria. Individuals could therefore benefit from these safe and effective dietary interventions to maintain the healthy gut bacteria and overall health. This study is being carried out to establish the effect of one such prebiotic, called galactooligosaccharide (B-GOS) on the relative balance of gut bacteria and metabolites in children with ASD. The aim is to enrol 42 children, ages 5-10 with formal ASD diagnosis and with signed informed consent from their parents, into double-blind, placebo controlled, parallel study. The trial will last 10 weeks in total (2 weeks run in period, 6 weeks treatment and 2 weeks follow up). Children will be required to take food supplement daily during the treatment period and their parents will collect stool, saliva and urine samples. Various questionnaires will also be used for assessments. Children will not be required to make other extra changes to their diet, medication or lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* children aged 5-10 years with formal ASD diagnosis
* children's parent or guardian has given written informed consent to participate and is willing to participate in the entire study

Exclusion Criteria:

* consumption of antibiotics, prebiotic or probiotics in the last 4 weeks prior to or during the study
* participants who have received bowel preparation for investigative procedures in the 4 weeks prior to the study
* undergone surgical resection of any part of the bowel

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
effect on faecal microbiota composition using pyrosequencing | change from baseline in microbiota composition to the end of treatment (6 months)
  using pyrosequencing
effect on faecal microbiota activity using nuclear magnetic resonance spectroscopy | change from baseline in microbiota activity to the end of treatment (6 months)
  using nuclear magnetic resonance spectroscopy

SECONDARY OUTCOMES:
questionnaire as a measure of bowel function | measured weekly for 6 months
  using weekly scores on questions related to stool consistency, frequency, abdominal pain and bloating
questionnaire as a measure of mood | monthly for 6 months
  using monthly scores on questions related to mood and sleep patterns
questionnaire as a measure of behaviour | monthly for 6 months
  using monthly scores on questions related to behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Jelena Vulevic, phd, Study Chair — Clasado Research Services
Locations (1):
- University of Reading, Reading, Berks, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
upon completion of the whole study, volunteers will be able to access their individual data following written request

REFERENCES:
- [Derived] Grimaldi R, Gibson GR, Vulevic J, Giallourou N, Castro-Mejia JL, Hansen LH, Leigh Gibson E, Nielsen DS, Costabile A. A prebiotic intervention study in children with autism spectrum disorders (ASDs). Microbiome. 2018 Aug 2;6(1):133. doi: 10.1186/s40168-018-0523-3. PMID 30071894